CLINICAL TRIAL: NCT01550770
Title: An Open Label, Exploratory Study of Propofol and Fentanyl Pharmacodynamics
Brief Title: Exploratory Study of Propofol and Fentanyl Pharmacodynamics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CI-10-0005
Record Dates: First submitted 2012-03-05; First posted 2012-03-12 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: General Anesthesia
MeSH Terms: interventions — Propofol

ARMS (1):
- proprofol (Experimental)
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — peripheral IV of propofol at increasing dose levels

SUMMARY:
Exploration of the hypothesis that general anesthesia is not a singular threshold but is a continuum of central nervous system depression dependent on interpretation of nociceptive stimuli.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesia (ASA) classification score I-II male and female volunteers
* Normal healthy individual by medical history and physical examination
* Uncomplicated airway anatomy
* Body Mass Index (BMI) between 18-29
* Subject willing to give consent and comply with evaluation and treatment schedule
* 18-55 years of age (inclusive)
* Negative durg screen for marijuana, cocaine, ecstasy, phencyclidine (PCP), amphetamines, benzodiazepines, opiates and methamphetamines
* Woman of childbearing age byst be utilizing reliable means of contraception
* Able to read, speak and understand English

Exclusion Criteria:

* Physical of psychological condition which would impair study participation as determined by the principal investigator
* Known or suspected neurological pathologies as assessed by the principal investigator
* History of significant alcohol or drug abuse, a history of allergy to opioids or propofol, or a history of chronic drug requirement or medical illness that is known to alter pharmacokinetics or pharmacodynamics of fentanyl and/or propofol
* Known or suspected hypersensitivity to any study drug
* Taken any medication within 2 days prior to study drug administration, with the exception of oral contraceptives
* Baseline tolerance above 50 mA on TES
* Pregnancy or lactation
* Consumed food within 8 hours or liquids within 4 hours prior to study drug administration
* Participation in any other investigational device or durg study within 30 days of enrollment
* Diagnosis of sleep apnea
* Current prescription to anti-depressant or anti-anxiety medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Difference between Modified Observers Assessment of Alertness (MOAAS) and transdermal electrical stimulation (TES) | 1 day
  MOAAS and TES assessment of increasing level(s) of sedation

CONTACTS AND LOCATIONS:
Overall Officials: Talmage Egan, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States